CLINICAL TRIAL: NCT03738748
Title: Effectiveness of the Ecoguided Percutaneous Neuromodulation of the Multipurpose Musculature of L-3 in Non-specific Chronic Lumbar Pain.
Brief Title: Effectiveness of Ecoguided Percutaneous Neuromodulation of the Multipurpose Musculature of L-3 in Non-specific Chronic Lumbar Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLA-12
Record Dates: First submitted 2018-10-20; First posted 2018-11-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: Neuromodulation; Low back pain; Ultrasound-guied percutaneous; TENS; Randomized Controlled Trial; Percutaneous stimulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided Percutaneous Neuromodulation (Experimental): This group will be treated with percutaneous neuromodulation using a needle with Physio Invasive® device, in its modality of percutaneous electrostimulation for 15 minutes, and guided by ultrasound equipment in the multifidus muscles of L3 (1 times/ 4 weeks).
  Interventions: Other: Ultrasound- guided Percutaneous Neuromulation
- TENS therapy (Active Comparator): The control group will apply a transcutaneous treatment with surface electrodes with TENS current at 170 Hz for 15 minutes in the L-3 region (1 times/ 4 weeks).
  Interventions: Other: TENS Therapy

INTERVENTIONS:
Other: Ultrasound- guided Percutaneous Neuromulation — The experimental group will be treated with percutaneous neuromodulation using a needle with Physio Invasive® device, in its modality of percutaneous electrostimulation for 15 minutes, and guided by ultrasound equipment in the multifidus muscles of L-3, once a week for 4 weeks.
  Arms: Ultrasound-guided Percutaneous Neuromodulation
Other: TENS Therapy — The control group will apply a transcutaneous treatment with surface electrodes with TENS current at 170 Hz for 15 minutes in the L-3 region, once a week for 4 weeks.
  Arms: TENS therapy

SUMMARY:
The study evaluates the effectiveness of Ultrasound-guided Percutaneous Neuromodulation in the lumbar multifidus of L3 in non-specific chronic low back pain.

DETAILED DESCRIPTION:
The effectiveness of neuromoduation in analgesic therapies has been more than contrasted. Considering that multifidus muscles, composed of the spinous transverse rotators muscles and spinous transverse multifidus muscles, are fundamental both for the static and for the dynamics of the lumbar spine, particularly for the region of L-3, the treatment of this musculature with ultrasound-guided percutaneous neuromodulation in patients with nonspecific chronic low back pain must have an analgesic repercussion in this nociceptive process.

Therefore, given that neuromodulation has been considered as a more than effective treatment in painful symptomatology and that diverse scientific literature has proven the activity of the multifida musculature directly affects the stability and mobility of the lumbar spine, it is more than likely interventions with neuromodulative treatments in the multifidus musculature at the level of the third lumbar vertebrae have positive results in Non-specific Chronic Low Back Pain.

ELIGIBILITY:
Inclusion Criteria:

* Score ≥4 on the Roland Morris Disability Questionnaire.
* Low back pain for ≥3 months
* Age between 18 and 65 years
* Not undergoing another physical therapy treatment

Exclusion Criteria:

* Presence of lumbar stenosis
* Diagnosis of spondylolisthesis
* Diagnosis of fibromyalgia
* Treatment with corticosteroid or oral medication within the past two weeks
* A history of spinal surgery
* Contraindication of analgesic electrical therapy
* Having previously received a treatment of electrical analgesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ) | At baseline and at 4 weeks (immediate post-treatment)
  This is a self-reported questionnaire consisting in 24 ítems reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Index (ODI). | At baseline and at 4 weeks (immediate post-treatment)
  It has 10 items associated to activities of daily living, each item has a puntuation fron 0 to 5 points.
Change from baseline in pain intensity (Visual Analogue Scale). | At baseline and at 4 weeks (immediate post-treatment)
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain.
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline and at 4 weeks (immediate post-treatment)
  It is a 17-item questionnaire that measures the fear of movement and (re)injury
Change from baseline on Quality of Life. | At baseline and at 4 weeks (immediate post-treatment)
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test | At baseline and at 4 weeks (immediate post-treatment)
  It measures the isometric endurance of trunk flexion muscles
Change from baseline in lumbar mobility flexion | At baseline and at 4 weeks (immediate post-treatment)
  It is determined by measuring the finger-to-floor distance
Change from baseline in range of motion and lumbar segmental mobility | At baseline and at 4 weeks (immediate post-treatment)
  This variable is quantified using the SpinalMouse® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagital spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

REFERENCES:
- [Background] Goubert D, De Pauw R, Meeus M, Willems T, Cagnie B, Schouppe S, Van Oosterwijck J, Dhondt E, Danneels L. Lumbar muscle structure and function in chronic versus recurrent low back pain: a cross-sectional study. Spine J. 2017 Sep;17(9):1285-1296. doi: 10.1016/j.spinee.2017.04.025. Epub 2017 Apr 26. PMID 28456669
- [Background] Freeman MD, Woodham MA, Woodham AW. The role of the lumbar multifidus in chronic low back pain: a review. PM R. 2010 Feb;2(2):142-6; quiz 1 p following 167. doi: 10.1016/j.pmrj.2009.11.006. PMID 20193941
- [Background] Rajfur J, Pasternok M, Rajfur K, Walewicz K, Fras B, Bolach B, Dymarek R, Rosinczuk J, Halski T, Taradaj J. Efficacy of Selected Electrical Therapies on Chronic Low Back Pain: A Comparative Clinical Pilot Study. Med Sci Monit. 2017 Jan 7;23:85-100. doi: 10.12659/msm.899461. PMID 28062862
- [Background] Bredow J, Bloess K, Oppermann J, Boese CK, Lohrer L, Eysel P. [Conservative treatment of nonspecific, chronic low back pain : Evidence of the efficacy - a systematic literature review]. Orthopade. 2016 Jul;45(7):573-8. doi: 10.1007/s00132-016-3248-7. German. PMID 27075679
- [Background] Wallwork TL, Stanton WR, Freke M, Hides JA. The effect of chronic low back pain on size and contraction of the lumbar multifidus muscle. Man Ther. 2009 Oct;14(5):496-500. doi: 10.1016/j.math.2008.09.006. Epub 2008 Nov 21. PMID 19027343
- [Background] Hides JA, Stanton WR, McMahon S, Sims K, Richardson CA. Effect of stabilization training on multifidus muscle cross-sectional area among young elite cricketers with low back pain. J Orthop Sports Phys Ther. 2008 Mar;38(3):101-8. doi: 10.2519/jospt.2008.2658. Epub 2007 Dec 7. PMID 18349481
- [Background] Kirby CC. A look at radiologic technology education. Radiol Technol. 1975 Sep-Oct;47(2):82-9. PMID 1188084
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692
- [Background] Nayak R, Banik RK. Current Innovations in Peripheral Nerve Stimulation. Pain Res Treat. 2018 Sep 13;2018:9091216. doi: 10.1155/2018/9091216. eCollection 2018. PMID 30302288
- [Background] Ilfeld BM, Gabriel RA, Said ET, Monahan AM, Sztain JF, Abramson WB, Khatibi B, Finneran JJ 4th, Jaeger PT, Schwartz AK, Ahmed SS. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Sciatic Nerve for Postoperative Analgesia Following Ambulatory Foot Surgery, a Proof-of-Concept Study. Reg Anesth Pain Med. 2018 Aug;43(6):580-589. doi: 10.1097/AAP.0000000000000819. PMID 29905630
- [Background] Ilfeld BM, Said ET, Finneran JJ 4th, Sztain JF, Abramson WB, Gabriel RA, Khatibi B, Swisher MW, Jaeger P, Covey DC, Robertson CM. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Femoral Nerve for Postoperative Analgesia Following Ambulatory Anterior Cruciate Ligament Reconstruction: A Proof of Concept Study. Neuromodulation. 2019 Jul;22(5):621-629. doi: 10.1111/ner.12851. Epub 2018 Aug 30. PMID 30160335
- [Background] Facci LM, Nowotny JP, Tormem F, Trevisani VF. Effects of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IFC) in patients with nonspecific chronic low back pain: randomized clinical trial. Sao Paulo Med J. 2011;129(4):206-16. doi: 10.1590/s1516-31802011000400003. PMID 21971895
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Gofeld M. Ultrasound-guided caudad epidural access for the lumbosacral neurostimulation: case report and technical note. Neuromodulation. 2011 Jan;14(1):68-71; discussion 71. doi: 10.1111/j.1525-1403.2010.00297.x. Epub 2010 Oct 7. PMID 21992165
- See also: Neuromodulación eléctrica y dolor raquídeo. — http://dx.doi.org/10.4321/S1134-80462015000300006
- See also: Spinal cord stimulation versus conventional medical management for neuropathic pain: A multicentre randomised controlled trial in patients with failed back surgery syndrome. — https://doi.org/10.1016/j.pain.2007.07.028
- See also: Prospective, Two-part Study of the Interaction Between Spinal Cord Stimulation and Peripheral Nerve Field Stimulation in Patients with Low Back Pain: Development of a New Spinal-Peripheral Neurostimulation Method — https://doi.org/10.1111/j.1525-1403.2010.00316.x